CLINICAL TRIAL: NCT07248995
Title: The Contribution of the Combination of Transthoracic and Transcranial Ultrasonography to the Titration of Positive End-expiratory Pressure in Patients With Acute Respiratory Distress Syndrome and Acute Brain Injury
Brief Title: Contribution of Transthoracic and Transcranial Ultrasonography to the Titration of PEEP in Patients With ARDS and ABI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Theodoros Schizodimos (Other)
Responsible Party: Sponsor-Investigator, Theodoros Schizodimos, Theodoros Schizodimos, George Papanicolaou Hospital
Organization: George Papanicolaou Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10957
Record Dates: First submitted 2025-11-14; First posted 2025-11-25 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Acute Respiratory Distress Syndrome (ARDS); Acute Brain Injury
MeSH Terms: conditions — Respiratory Distress Syndrome; Brain Injuries | interventions — Positive-Pressure Respiration

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stepwise PEEP Elevation Protocol Arm (Experimental): All participants with ARDS and ABI will undergo a protocolized stepwise increase of PEEP at four levels. Each participant will serve as their own control.
  Interventions: Procedure: Stepwise Positive End-Expiratory Pressure (PEEP) Increase Protocol

INTERVENTIONS:
Procedure: Stepwise Positive End-Expiratory Pressure (PEEP) Increase Protocol — The intervention includes a stepwise increase in PEEP level from 5 to 8, 12 and 16 centimeter of water (cmH2O). After each PEEP level change, lung ultrasound and transcranial doppler will be performed, and the values of intracranial pressure (ICP) and brain oxygen partial pressure (PO2), as well as the mechanical ventilation parameters, will be recorded. Arterial blood gases will be taken 20 minutes later.

SUMMARY:
The present study will investigate whether the combined use of lung and brain ultrasonography is useful in selecting the optimal positive end-expiratory pressure in mechanically ventilated critically ill patients with acute respiratory distress syndrome and acute brain injury, aiming at an individualized, brain-protective ventilation strategy.

DETAILED DESCRIPTION:
The present study aims to evaluate whether the combined use of lung ultrasonography and brain ultrasonography can assist in determining the optimal positive end-expiratory pressure (PEEP) in mechanically ventilated, critically ill patients with acute respiratory distress syndrome (ARDS) and acute brain injury (ABI). In patients with concomitant respiratory and neurological injury, selecting an appropriate PEEP level is particularly challenging, as strategies that improve lung aeration may simultaneously increase intracranial pressure or compromise cerebral hemodynamics.

Lung ultrasound will be used to assess aeration patterns and guide lung recruitment through the Lung Ultrasound Score (LUS), while transcranial Doppler ultrasonography will be used to evaluate cerebral blood flow and intracranial pressure surrogates, such as the pulsatility index. By integrating both assessments, the study seeks to identify a PEEP level that optimizes pulmonary function while minimizing adverse effects on cerebral physiology. The overarching goal is to develop an individualized, brain-protective ventilation strategy for patients with ARDS and ABI.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Severe acute brain injury (e.g., traumatic brain injury, subarachnoid hemorrhage, intracerebral hemorrhage, acute ischemic stroke)
* Development of ARDS (according to Berlin criteria) within the first 10 days of ICU admission

Exclusion Criteria:

* Severe chronic brain diseases
* Brain tumor or central nervous system (CNS) infection
* Severe chronic pulmonary or cardiovascular disease
* Severe coagulopathy
* Undergoing decompressive craniectomy
* Lack of invasive neuromonitoring
* Withdrawal of life-sustaining treatment
* Poor acoustic window in ultrasound

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Difference in PEEP Levels Between Optimal PEEP (LUS-Guided) and Safe PEEP (TCD and Respiratory Mechanics-Guided) | From the start of the intervention until completion of the PEEP titration procedure, within approximately 120 minutes from intervention initiation.
  Optimal PEEP is determined using the Lung Ultrasound Score (LUS; aeration score 0-36), while Safe PEEP is determined based on Transcranial Doppler (TCD) measurements (Pulsatility Index, mean flow velocity) and respiratory mechanics parameters (driving pressure, plateau pressure, compliance). The outcome represents the difference between Optimal PEEP and Safe PEEP expressed in cmH₂O.
  Unit of Measure: cmH₂O

SECONDARY OUTCOMES:
Correlation Between PEEP Difference and Clinical Outcomes | From the intervention until ICU discharge and hospital discharge, assessed up to 90 days
  Correlation between the difference in PEEP levels (cmH₂O) and the following clinical outcomes: duration of mechanical ventilation, ICU length of stay, and ICU/hospital mortality.
  Unit of Measure:
  PEEP difference: cmH₂O, Duration of mechanical ventilation: days, ICU length of stay: days, ICU mortality: %, Hospital mortality: %

CONTACTS AND LOCATIONS:
Overall Officials: Theodoros Schizodimos, MD, Principal Investigator — 2nd Intensive Care Unit, George Papanikolaou General Hospital of Thessaloniki
Locations (1):
- George Papanikolaou General Hospital, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2025-10-19): https://cdn.clinicaltrials.gov/large-docs/95/NCT07248995/Prot_000.pdf
  • Statistical Analysis Plan (2025-10-19): https://cdn.clinicaltrials.gov/large-docs/95/NCT07248995/SAP_001.pdf